CLINICAL TRIAL: NCT02856386
Title: Assessment of the Utility of a Dietary Supplement as an Adjunct to Standard of Care for Children With Chronic Diarrhea
Brief Title: Use of a Dietary Supplement to Support Digestive Health in Children With Chronic Diarrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LiveLeaf Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-001
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Antibiotic-associated Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- polyphenol supplement (Experimental): Dietary supplement administered 8 mL once daily
  Interventions: Dietary Supplement: polyphenol supplement

INTERVENTIONS:
Dietary Supplement: polyphenol supplement — 8 mL once daily
  Other Names: Traveler Protect

SUMMARY:
Micronutrients missing in the diet may assist in supporting digestive health in children with chronic GI issues. This study will monitor changes in symptoms associated with digestive problems in children provided with a dietary supplement that will be taken in conjunction with the standard of care.

DETAILED DESCRIPTION:
Children with GI symptoms have varying response to the standard of care treatments. A dietary supplement of polyphenols from green tea and pomegranate extracts provides micronutrients often missing from conventional American diets. The objective of this study is to monitor changes in GI symptoms when the supplement is provided alongside the standard of care for children with symptoms that have been present for more than two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients with diagnosis of unresolved gastrointestinal distress
* Parent or guardian willing to administer the dietary supplement orally once daily for up to 21 days
* Parent or guardian willing to record changes in GI symptoms on a questionnaire
* Parent or guardian willing to bring the child for a clinic visit to close-out participation in the study

Exclusion Criteria:

* requires care in an ICU
* has documented intestinal stricture, stenosis, obstruction, or abscess
* has concomitant congenital diseases
* are immunodeficient
* has malformation of the GI tract
* is unable to swallow fluids
* parent or guardian is unable or unwilling to provide informed consent

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of GI symptoms | 3 weeks

IPD SHARING:
Plan to Share IPD: No